CLINICAL TRIAL: NCT02471651
Title: Dexamethasone Intravitreal Implant (0.7mg) for the Treatment of Persistent Diabetic Macular Edema Following Intravitreal Anti-Vascular Endothelial Growth Factor Therapy
Brief Title: Dexamethasone Intravitreal Implant for the Treatment of Persistent Diabetic Macular Edema
Acronym: DIME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: California Retina Consultants (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC2015-02
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Ranibizumab; Bevacizumab; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implant (Active Comparator): Subjects randomized to dexamethasone intravitreal implant (0.7mg) will receive the initial treatment at Month 3 (visit 4) and Month 6 (visit 7) and are eligible to receive one additional dose at Month 9 (visit 10), Month 10 (visit 11) or Month 11 (visit 12) for persistent or recurrent macular edema documented on SDOCT. If dexamethasone intravitreal implant (0.7mg) is administered at Month 10 (visit 11) or Month 11 (visit 12) an additional safety study visit will be required at one to two months following Month 12 (visit 13). The investigator can withhold treatment with dexamethasone intravitreal implant (0.7mg) beginning at Month 9 if there is complete resolution of diabetic macular edema document on SDOCT.
  Interventions: Drug: Dexamethasone intravitreal implant (0.7 mg)
- Intravitreal anti-VEGF injection (Active Comparator): Subjects randomized to continue on anti-vegf therapy will receive intravitreal anti-vegf injections at Month 3 (visit 4) Month 4 (visit 5) and Month 5 (visit 6). Beginning at Month 6 (visit 7), subjects who have received 6 intravitreal anti-vegf injections and continue to present with persistent diabetic macular edema defined as less than 10% reduction or any increase in CST compared to baseline values and CST is greater than 300 microns, will receive dexamethasone intravitreal implant (0.7mg) at Month 6 (visit 7) and Month 9 (visit 10). The follow-up period for all subjects will continue through 12 months from the baseline study visit.
  Interventions: Drug: Intravitreal anti-VEGF injection

INTERVENTIONS:
Drug: Dexamethasone intravitreal implant (0.7 mg) — Subjects with persistent DME who are randomized to this arm may get up to 3 treatments with the implant (0.7 mg dexamethasone).
  Other Names: Ozurdex
  Arms: Implant
Drug: Intravitreal anti-VEGF injection — This injection may be ranibizumab, bevacizumab, or aflibercept.
  Other Names: ranibizumab, bevacizumab, or aflibercept
  Arms: Intravitreal anti-VEGF injection

SUMMARY:
Laser photocoagulation and intravitreal anti-vascular growth factor injections are commonly used treatment options for individuals with diabetic macular edema. However, some patients continue to experience persistent diabetic macular edema and poor vision despite continued laser and/or anti-vegf therapy. Recent clinical trials suggest that due to inflammatory mediators dexamethasone intravitreal implant (0.7mg) may be a good alternative therapy for individuals unresponsive to laser photocoagulation or intravitreal anti-vascular growth factor injections. The purpose of this research study is to compare the effectiveness of using a dexamethasone steroid implant versus monthly intravitreal anti-VEGF injections for research participants with persistent diabetic macular edema (DME).

DETAILED DESCRIPTION:
Macular edema is a major cause of central vision loss in patients presenting with diabetic retinopathy. Diabetic macular edema (DME) occurs when fluid leaks into the center of the macula, the part of the eye where sharp, straight-ahead vision occurs. The fluid makes the macula swell, blurring vision. Diabetic macular edema (DME) affects between 8% to 10% of 23.6 million diabetic individuals in the United States. The prevalence of diabetic macular edema after 15 years of known diabetes is approximately 20% in patients with type 1 diabetes, 25% in patients with type 2 diabetes who are taking insulin, and 14% in patients with type 2 diabetes who do not take insulin. Within two years of diagnosis, nearly half of individuals with DME will lose 2 or more lines of visual acuity (the smallest line you can read on a standardized vision chart held 20 feet away).

Diabetic macular edema is typically treated with laser and/or intravitreal injections of drugs such as anti-VEGF agents. Anti-VEGF agents block a protein that slows the growth of the abnormal blood vessels. Dexamethasone is a corticosteroid used to treat inflammation. Dexamethasone implant is a steroid implant injected into the eye to treat swelling that may occur when there is a blockage of certain blood vessels in your eyes. Both anti-VEGF agents and dexamethasone implant are approved by the FDA to treat DME.

The purpose of this research study is to compare the effectiveness of using a dexamethasone steroid implant versus monthly intravitreal anti-VEGF injections for research participants with persistent diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and comply with study assessments for the full duration of the study.
* Age ≥ 18 years
* Diagnosis of diabetes mellitus (type 1 or 2)

  * Any one of the following will be considered to be sufficient evidence that diabetes is present:
  * Current regular use of insulin for treatment of diabetes
  * Current regular use of oral anti-hyperglycemia agent for the treatment of diabetes
* Clinical evidence of retinal thickening due to macular edema involving the center of the macula associated with diabetic retinopathy.
* Previous history of anti-vegf treatment for diabetic macular edema (DME) with documented incomplete resolution of central subfield thickening by spectral-domain optical coherence tomography (SDOCT). At least 4 intravitreal anti-vegf injections within the past six months prior to the baseline study visit are required for eligibility.
* Central diabetic macular edema present on clinical examination and SDOCT testing with central 1 mm subfield thickness greater than 300 microns as measured on SDOCT at the baseline visit.
* Visual acuity score greater than or equal to 19 letters (20/400) and less than or equal to 74 letters (20/32) by the ETDRS visual acuity protocol.
* Media clarity, pupillary dilation and patient cooperation sufficient to allow SDOCT testing and retinal photography.

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or known to be pregnant; also pre-menopausal women not using adequate contraception.
* Participation in another ocular investigation or trial simultaneously
* Blood pressure > 180/110 mmHg (systolic above 180 OR diastolic above 110 mmHg)
* Any condition that, in the opinion of the investigator, would preclude participation in the study (e.g. chronic alcoholism, drug abuse)
* Evidence of vitreoretinal interface abnormality after ocular exam or OCT that may be contributing to the macular edema
* An eye that, in the investigator's opinion, has no chance of improving in visual acuity following resolution of macular edema (e.g. presence of subretinal fibrosis or geographic atrophy)
* Presence of another ocular condition that may affect the visual acuity or macular edema during the course of the study (e.g. AMD, uveitis, Irvine-Gass)
* Evidence of active neovascularization of the iris or retina
* Evidence of central atrophy or fibrosis in the study eye
* Presence of substantial cataract, one that might decrease the vision by 3 or more lines of vision at sometime during the study.
* History of vitreous surgery in the study eye
* History of cataract surgery within 3 months of enrollment.
* History of YAG capsulotomy within 2 months of enrollment.
* Visual acuity <20/400 on ETDRS visual acuity charts in the fellow eye
* Uncontrolled glaucoma (pressure > 30 mmHg) despite treatment with glaucoma medications.
* History of cerebral vascular accident or myocardial infarction within 3 months prior to Day 0.
* Use of systemic steroids (eg, oral, intravenous, intramuscular, epidural, rectal, or extensive dermal) within one month prior to the baseline study visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Gordon, Ph.D., Study Director — California Retina Consultants
Locations (4):
- United States (4):
  - California Retina Consultants, Bakersfield, California
  - California Retina Consultants, Oxnard, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants, Santa Maria, California

REFERENCES:
- [Derived] Chakravarthy H, Devanathan V. Molecular Mechanisms Mediating Diabetic Retinal Neurodegeneration: Potential Research Avenues and Therapeutic Targets. J Mol Neurosci. 2018 Nov;66(3):445-461. doi: 10.1007/s12031-018-1188-x. Epub 2018 Oct 6. PMID 30293228

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Implant | Intravitreal Anti-VEGF Injection
Started | 20 | 20
Completed | 15 | 15
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Implant | Intravitreal Anti-VEGF Injection | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age assessment was done for subjects who completed the study; subjects who were dropped from the study prior to their month 12 visit were not analyzed.
  years
    number analyzed (Participants) | 15 | 15 | 30
    (all) | 62 (8) | 65 (7) | 63 (8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender assessment was done for subjects who completed the study; subjects who were dropped from the study prior to their month 12 visit were not analyzed.
  Participants
    number analyzed (Participants) | 15 | 15 | 30
    Female | 7 | 8 | 15
    Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Assessments were done for subjects who completed the study; subjects who were dropped from the study prior to their month 12 visit were not analyzed.
  Participants
    number analyzed (Participants) | 15 | 15 | 30
    Hispanic or Latino | 7 | 7 | 14
    Not Hispanic or Latino | 8 | 8 | 16
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Assessments were done for subjects who completed the study; subjects who were dropped from the study prior to their month 12 visit were not analyzed.
  Participants
    number analyzed (Participants) | 15 | 15 | 30
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 0 | 0 | 0
    White | 14 | 15 | 29
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: Assessments were done for subjects who completed the study; subjects who were dropped from the study prior to their month 12 visit were not analyzed.
  participants
    United States: number analyzed (Participants) | 15 | 15 | 30
    United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Central 1 mm Subfield Thickness Between Baseline and 9 Months
Description: Mean change in central 1 mm sub-field thickness between baseline and 9 months as measured by Spectral Domain Optical Coherence Tomography (SDOCT).
Time Frame: baseline and 9 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Implant | Intravitreal Anti-VEGF Injection
Number analyzed (Participants) | 15 | 15
millimeters | -51 (117) | -60 (149)

2. Secondary Outcome: Mean Change in Standardized Best-corrected Visual Acuity (BCVA) Between Baseline and 9 Months
Description: Mean change in standardized best-corrected visual acuity between baseline and 9 months as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) testing. Participants were challenged with reading letters on lines of an eye chart (5 letters per line). Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until they reached a row where a minimum of three letters on a line could be read, and were scored by how many letters could be correctly identified
Time Frame: baseline and 9 months
Measure: Mean (Standard Deviation); unit: letters on the ETDRS scale
Arm/Group | Implant | Intravitreal Anti-VEGF Injection
Number analyzed (Participants) | 15 | 15
letters on the ETDRS scale | 1.5 (13) | 1.8 (12)

3. Secondary Outcome: Total Number of Treatments in Each Arm Between Baseline and 9 Months
Description: Total number of treatments in each arm between baseline and 9 months.
Time Frame: baseline and 9 months
Measure: Number; unit: injections
Arm/Group | Implant | Intravitreal Anti-VEGF Injection
Number analyzed (Participants) | 15 | 15
injections | 43 | 83

ADVERSE EVENTS:
Time Frame: 12 months.
Description: AEs and SAEs were monitored at every visit and recorded.
Arm/Group | Implant | Intravitreal Anti-VEGF Injection
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20
Other Adverse Events (participants affected / at risk) | 10/20 | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implant (N=20) | Intravitreal Anti-VEGF Injection (N=20)
Skin graft (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin Graft (Leg, R)
Rhegmatogenous Retinal Detachment (Eye disorders) | 0 (0) | 1 (1) — Rhegmatogenous Retinal Detachment in study eye
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implant (N=20) | Intravitreal Anti-VEGF Injection (N=20)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pinched Nerve (Nervous system disorders) | 0 (0) | 1 (1)
tooth ache (General disorders) | 0 (0) | 1 (1)
High IOP (Eye disorders) | 4 (5) | 1 (1)
Eye Pain (Eye disorders) | 1 (1) | 2 (2)
active neovascularization (Eye disorders) | 0 (0) | 1 (1)
flu (General disorders) | 0 (0) | 2 (3)
hypertension (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Continuing/increased macular edema (Vascular disorders) | 0 (0) | 1 (3)
subconjunctival irritation (Eye disorders) | 0 (0) | 1 (1)
vitreous hemorrhage (Vascular disorders) | 0 (0) | 1 (2)
tooth being pulled (General disorders) | 0 (0) | 1 (1)
cold/cough (General disorders) | 4 (6) | 0 (0)
iron deficiency (General disorders) | 1 (1) | 0 (0)
headache (General disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
viral conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
leg injury (General disorders) | 1 (1) | 0 (0) — leg injury due to fall
eye itchiness (Eye disorders) | 1 (1) | 0 (0)
Toe infection (Infections and infestations) | 1 (1) | 0 (0)
dry eye (Eye disorders) | 0 (0) | 1 (1)
general fatigue (General disorders) | 0 (0) | 1 (1)
stomach virus (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT02471651/Prot_SAP_000.pdf